CLINICAL TRIAL: NCT06034769
Title: Oral Health, Temporomandibular Dysfunction and Oropharyngeal Dysphagia in Bipolar Patients
Brief Title: Oral and Jaw Health in Bipolar Patients
Status: Completed | Type: Observational
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Hazel Çelik Güzel, Assist. Prof. Dr, Bandırma Onyedi Eylül University
Other Study IDs: 2023-44
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Bipolar Disorders; Oral Health
Keywords: Bipolar disorders; Oral health; Temporomandibular disorders
MeSH Terms: conditions — Bipolar Disorder; Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The assessment of oral health, jaw health and related problems in bipolar patients is important to provide a holistic approach to patients in terms of physical, mental and psychosocial aspects and to improve quality of life. In this study, oral health, temporomandibular dysfunction (TMD) and oropharyngeal dysphagia (OD) were investigated in patients with Bipolar Disorder (BD).

DETAILED DESCRIPTION:
During the remission period, 70 individuals aged 20-60 years with BD were divided into two groups according to the duration of diagnosis as under ten years (Group 1=33) and over ten years (Group 2=37). Oral and dental health-related quality of life was assessed with the Oral Health Impact Profile-14 (OHIP-14), TMJ pain was assessed with the Numeric Pain Scale (NPS), the presence of TMJ discomfort was assessed with the Fonseca Anamnestic Questionnaire (FAQ), chewing functionality was assessed with the Jaw Function Limitation Scale-8 (JFLS-8), and oropharyngeal dysphagia was assessed with the Eating Assessment Tool (EAT-10).

ELIGIBILITY:
Inclusion Criteria:

* Patients between 20 and 60 years of age who volunteered to participate in the study and signed the informed consent form,
* diagnosed with BD at the outpatient department of Bakırkoy Prof. Dr. Mazhar Osman Mental Health and Neurological Diseases Training and Research Hospital,
* in remission for at least 3 months,
* had a history of regular lithium use for at least 1 year in any phase of the disease were included in the study.

Exclusion Criteria:

* being in a manic or depressive episode (Young Mania Rating Scale score greater than 7, Hamilton Depression Rating Scale score greater than 7)
* history of comorbid psychiatric illness,
* alcohol and substance use disorder,
* cancer, neurological problems, congenital anomalies, musculoskeletal problems, systemic illness,
* facial paralysis,
* spinal, abdominal and/or TMJ surgery,
* and having received any spinal or TMJ treatment in less than 6 months.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with bipolar disorder in remission
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Oral Health Impact Profile-14 (OHIP-14) | February 2023- July 2023
  This scale, which has been shown to be valid and reliable in measuring oral and dental health-related quality of life, consists of 14 questions in 7 dimensions. Each question is scored from 0 (never) to 4 (always). The scale ranges from 0 to 56, with high scores indicating poor quality of life.
Numerical Pain Scale (NPS) | February 2023- July 2023
  This simple, valid and reliable method, often used to measure pain intensity in the clinic, asks the participant to mark a number on a 10 cm scale with numbers ranging from '0' (no pain) to '10' (unbearable pain) for the pain felt in the TMJ region
Fonseca Anamnestic Questionnaire (FAQ) | February 2023- July 2023
  This scale, which has been shown to be valid and reliable as a TMD assessment tool, consists of 10 questions. A score of 25 or more on the scale indicates the presence of TMD.
Jaw Functional Limitation Scale-8 (JFLS-8) | February 2023- July 2023
  This scale, which has demonstrated validity and reliability, provides an assessment of chewing functionality during various activities of the jaw and consists of 8 questions. On this scale, which ranges from 0-80, a high score indicates limited chewing functionality.
Eating Assessment Tool (EAT-10) | February 2023- July 2023
  This scale, which assesses the symptoms and severity of oropharyngeal swallowing disorder and has been shown to be valid and reliable, consists of 10 questions. A total score of 3 and above on the scale, indicates the presence of a swallowing problem.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakırkoy Prof. Dr. Mazhar Osman Mental Health and Neurological Diseases Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided